CLINICAL TRIAL: NCT05987072
Title: A PHASE 1, OPEN-LABEL, SINGLE-ARM STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY, AND TOLERABILITY FOLLOWING SINGLE AND MULTIPLE DOSES OF SISUNATOVIR IN CHINESE HEALTHY PARTICIPANTS
Brief Title: A Study to Learn How the Study Medicine Called Sisunatovir is Tolerated and Acts in the Bodies of Chinese Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C5241018
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — sisunatovir

STUDY DESIGN:
Intervention Model Description: single-arm to investigate PK, safety and tolerability of 200 mg sisunatovir given as a single dose on Day 1 in a fasted state followed by repeated twice daily doses (200 mg BID, Q12 hours) from Days 4-7 plus 1 morning dose on Day 8 in a fed state in Chinese healthy participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): This only arm will be given as a single dose on Day 1 in a fasted state followed by repeated twice daily doses (200 mg BID, Q12 hours) from Days 4-7 plus 1 morning dose on Day 8 in a fed state
  Interventions: Drug: Sisunatovir

INTERVENTIONS:
Drug: Sisunatovir — Will be given as a single dose on Day 1 in a fasted state followed by repeated twice daily doses (200 mg BID, Q12 hours) from Days 4-7 plus 1 morning dose on Day 8 in a fed state

SUMMARY:
The purpose of the study is to learn about:

* The activity of sisunotavir in the body over a period. It includes the processes by which sisunotavir is absorbed, distributed in the body, localized in the tissues, and removed from the body.
* safety and tolerability of sisunatovir (PF-07923568) in Chinese healthy adult participants.

This information is being collected to support further clinical development as well as medicine registration in China.

This study is seeking for participants who:

* are male and female participants aged 18 to 65 years of age.
* are male and female participants who are healthy as seen by medical tests.
* have body mass index (BMI) of 19 to 27 kg/m2 and a total body weight of more than 50 kilograms (110 pounds).

About 12 participants will receive sisunatovir. Four capsules (strength=50 milligrams, 200 milligrams in total) of Sisunatovir will be given on Day 1 on empty stomach. This will be followed by 8 capsules of sisunatovir with 12 hours gap in between four capsules from Days 4 to 7. The participants will have to take 4 capsules of sisunatovir in the morning of 8th day with a meal.

The total time of participants will be in the study is about 71 days. This includes the screening visit to the Follow-up contact. In screening visit, participants will be tested to see if they are fit to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male and female participants aged 18 to 65 years of age, inclusive, at the time of signing of the informed consent document (ICD).
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, standard 12-lead ECG, and laboratory tests.
* Body mass index (BMI) of 19 to 27 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality, or other conditions or situations related to coronavirus disease 2019 (COVID-19) pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention with the exception of moderate/strong cytochrome P4503A (CYP3A) inducers or time-dependent inhibitors which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
* A positive urine drug test, confirmed by a repeat test, if deemed necessary.
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTc corrected using Fridericia's formula [QTcF] >450 ms, complete left bundle branch block [LBBB], signs of an acute or indeterminate- age myocardial infarction, ST-segment and T-wave [ST-T] interval changes suggestive of myocardial ischemia, second- or thirddegree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate-corrected using the Fridericia method only and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 ms, or quantitative restrictions (QRS) exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer interpreted- ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:
* Glomerular filtration rate (GFR) <60 mL/min/1.73m2 based on chronic kidney disease epidemiology (CKD-EPI equation);
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.05 × upper limit of normal (ULN);
* Gamma-glutamyl transferase (GGT) > 1.05 × ULN;
* Alkaline phosphatase > 1.05 × ULN;
* Total bilirubin level ≥1.05 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- China (3):
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve participants were enrolled and treated in the study.
Pre-assignment Details: Follow-up occurred via telephone contact and must occur 28 to 35 days after administration of the last dose of study intervention.
Groups:
- Sisunatovir 200 mg: Participants received a single oral dose of sisunatovir 200 mg on Day 1 in a fasted state followed by repeated twice daily doses (200 mg BID, every 12 hours [Q12 hours]) from Days 4-7 plus 1 morning dose on Day 8 in a fed state.
Period: Treatment Period (Day -1 to Day 11)
Arm/Group | Sisunatovir 200 mg
Started | 12
Received Treatment | 12
Completed | 12
Not Completed | 0
Period: FOLLOW-UP
Arm/Group | Sisunatovir 200 mg
Started | 12
Received Treatment | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was defined as all participants enrolled and who took at least 1 dose of study intervention.
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.4 (4.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sisunatovir on Day 1
Description: Cmax was defined as maximum observed plasma concentration. Cmax was observed directly from data.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72 hours post dose on Day1
Population: Analysis population included all participants who take at least 1 dose of study intervention and in whom at least 1 plasma concentration value is reported. One participant had emesis on Day 1 and therefore was excluded from the summaries.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 11
nanogram per milliliter (ng/mL) | 80.14 (73)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sisunatovir on Day 4
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12 hours post dose on Day 4
Population: Analysis population included all participants who take at least 1 dose of study intervention and in whom at least 1 plasma concentration value is reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
nanogram per milliliter (ng/mL) | 115.5 (59)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sisunatovir on Day 8
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72 hours post dose on Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
nanogram per milliliter (ng/mL) | 198.7 (51)

4. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time 12 Hours (AUC12) of Sisunatovir on Day 1
Description: AUC12 was defined as area under the concentration-time curve from time zero to 12 hours.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12 hours post dose on Day1
Population: Analysis population included all participants who take at least 1 dose of study intervention and have at least 1 of the PK parameters of interest calculated. One participant had emesis on Day 1 and therefore was excluded from the summaries.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 11
nanogram*hour per milliliter (ng*hr/mL) | 470.6 (71)

5. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time 12 Hours (AUC12) of Sisunatovir on Day 4
Description: AUC12 was defined as area under the concentration-time curve from time zero to 12 hours.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12 hours post dose on Day 4
Population: Analysis population included all participants who take at least 1 dose of study intervention and have at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
nanogram*hour per milliliter (ng*hr/mL) | 602.3 (60)

6. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time 12 Hours (AUC12) of Sisunatovir on Day 8
Description: AUC12 was defined as area under the concentration-time curve from time zero to 12 hours.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12 hours post dose on Day 8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
nanogram*hour per milliliter (ng*hr/mL) | 1295 (65)

7. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of Sisunatovir on Day1
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72 hours post dose on Day1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 11
nanogram*hour per milliliter (ng*hr/mL) | 708.8 (78)

8. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) on Day1
Description: AUCinf was defined as area under the concentration-time curve from time 0 to infinity.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72 hours post dose on Day1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 11
nanogram*hour per milliliter (ng*hr/mL) | 757.3 (70)

9. Secondary Outcome: Time to Reach Cmax (Tmax) on Day 1, Day 4 and Day 8
Description: Tmax was defined as time to reach Cmax.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72 hours post dose on Day1, and Day 8. 0, 1, 2, 3, 4, 5, 6, 8, 10, 12 hours post dose on Day 4.
Population: Analysis population included all participants who take at least 1 dose of study intervention and have at least 1 of the PK parameters of interest calculated. One participant had emesis on Day 1 and therefore was excluded from the summaries of Day 1.
Measure: Median (Full Range); unit: hr (hour)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
hr (hour)
  Day 1: number analyzed (Participants) | 11
  Day 1 | 5.00 [2.00 to 5.00]
  Day 4 | 5.00 [3.00 to 6.00]
  Day 8 | 5.00 [3.00 to 6.00]

10. Secondary Outcome: Terminal Elimination Half-life (t½) on Day 1 and Day 8
Description: t½ was defined as terminal elimination half-life.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12,14, 24, 48, 72 hours post dose on Day1, and Day 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hr (hour)
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
hr (hour)
  Day 1: number analyzed (Participants) | 11
  Day 1 | 9.495 (1.5588)
  Day 8 | 10.40 (1.2316)

11. Secondary Outcome: Accumulation Ratio for Sisunatovir (Rac)
Description: Rac is defined as: Observed accumulation ratio for AUCtau. Accumulation ratio on AUCtau = AUC12 (Day 8) /AUC12 (Day 4)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12 hours post dose on Day 4 and Day 8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
ratio | 2.149 (29)

12. Secondary Outcome: Accumulation Ratio on Cmax for Sisunatovir (Rac, Cmax)
Description: Accumulation ratio on Cmax =Cmax (Day 8) /Cmax (Day 4)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 10, 12 hours post dose on Day 4 and 0, 1, 2, 3, 4, 5, 6, 8, 10, 12,14, 24, 48, 72 hours post dose on Day 8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
ratio | 1.720 (26)

13. Secondary Outcome: Number of Participants With All-Causality and Treatment-Related Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship with the study intervention. SAE is defined as one of the following: is fatal or life threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; is medically significant; requires inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AE is defined as an AE with onset date occurring during the on-treatment period. AEs include all SAEs and non-SAEs.
Time Frame: From the first dose (Day 1) up to 35 days after the last dose (Day 8) of study intervention (up to 43 days)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
Participants
  Participants with all-causality TEAEs | 7
  Participants with all-causality SAEs | 0
  Participants with treatment related TEAEs | 6
  Participants with treatment related SAEs | 0

14. Secondary Outcome: Number of Participants With Vital Signs Meeting the Pre-specified Criteria
Description: Blood pressure (BP) and pulse rate were obtained with participant following at least a 5-minute rest in a supine position. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline up to Day 11 (11 days)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
Participants
  supine systolic BP value<90 mmHg | 0
  supine systolic BP increase≥ 30 mmHg | 0
  supine systolic BP decrease≥ 30 mmHg | 1
  supine diastolic BP value< 50mmHg | 0
  supine diastolic BP increase≥ 20mmHg | 0
  supine diastolic BP decrease≥ 20mmHg | 1
  pulse rate value<40 bpm | 0
  pulse rate value>120 bpm | 0

15. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, platelet, neutrophils, eosinophils, monocytes, basophils, lymphocytes, leukocytes); clinical chemistry (alanine aminotransferase, albumin, alkaline phosphatase, bilirubin, calcium, carbon dioxide combining power, chloride, creatinine, cystatin C, GFR CKD-EPI serum creatinine 2021, gamma glutamyl transferase, glucose, potassium, sodium, urate, urea). urinalysis (Bilirubin, Glucose, Hemoglobin, Ketones, Leukocyte Esterase, Nitrite, Protein, Urobilinogen, pH).0 indicates no participants with abnormalities of all above lab examination.
Time Frame: Baseline up to Day 11 (11 days)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
Participants | 0

16. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities: maximum PR interval >=300 milliseconds (msec) and maximum increase PR interval increase from baseline (IFB): percent change (Pctchg) >=25 percent (%) for baseline value of >200 msec and Pctchg>=50% for baseline value of <=200 msec for PR interval, maximum QRS interval >=140 msec and a maximum IFB: Pctchg>=50%, maximum QTCF interval (Fridericia's Correction) of 450 msec to <480 msec, 480 msec to <500 msec or >=500 msec and a maximum change of <=30change<60 or >=60 msec from baseline.
Time Frame: Baseline up to Day 11 (11 days)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 200 mg
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: From the first dose (Day 1) up to 35 days after the last dose (Day 8) of study intervention (up to 43 days)
Arm/Group | Sisunatovir 200 mg
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sisunatovir 200 mg (N=12)
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT05987072/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05987072/SAP_001.pdf